CLINICAL TRIAL: NCT02932735
Title: The Efficacy of Probe-based Confocal Laser Endomicroscopy in Staging OLGIM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of Qilu Hospital, Shandong University
Other Study IDs: 2016SDU-QILU-18
Record Dates: First submitted 2016-10-10; First posted 2016-10-13 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Probe-based Confocal Laser Endomicroscopy; the Operative Link on Gastric Intestinal Metaplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Gastric intestinal metaplasia (GIM) is an important premalignant lesion for gastric cancer. Precisely surveillance of patients with GIM may result in early detection and improved prognosis. Though important, it is not necessary to recommend surveillance endoscopy for all patients with GIM, since the progression rate to gastric cancer within 10 years is only 1.8% in those patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 40 years or older with Helicobacter pylori infection;
* Histologically verified GIM, atrophic gastritis or dysplasia.

Exclusion Criteria:

* Patients with gastrectomy, acute GI bleeding and advanced gastric cancer;
* Conditions unsuitable for performance of pCLE, such as coagulopathy, impaired renal function or allergy to fluorescein sodium;
* Pregnancy or breastfeeding;
* Inability to provide informed consent and other situations that could interfere with the examination or therapeutic protocol.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients scheduled for pCLE examination will be recruited in this study at Qilu Hospital, Shandong University.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
the sensitivity of probe-based Confocal Laser Endomicroscopy (pCLE) in staging the Operative Link on Gastric Intestinal Metaplasia (OLGIM). | 6 months
the of specificity of probe-based Confocal Laser Endomicroscopy (pCLE) in staging the Operative Link on Gastric Intestinal Metaplasia (OLGIM). | 6 months

SECONDARY OUTCOMES:
the of sensitivity of probe-based Confocal Laser Endomicroscopy (pCLE) in staging Gastric Intestinal Metaplasia (GIM). | 6 months
the of specificity of probe-based Confocal Laser Endomicroscopy (pCLE) in staging Gastric Intestinal Metaplasia (GIM). | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Li Yanqing, MD, PhD, Principal Investigator — Qilu Hospital of Shandong University

IPD SHARING:
Plan to Share IPD: No